CLINICAL TRIAL: NCT04063787
Title: Use of an Intermittent Pneumatic Compression Device to Promote Vein Dilation in Patients With Kidney Disease to Enable Creation of Arteriovenous Fistulas
Brief Title: Intermittent Pneumatic Compression Device for Vein Dilation in Kidney Disease Patients to Enable AVF Creation (FACT)
Acronym: FACT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: Fist Assist Devices, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB19-0306
Record Dates: First submitted 2019-08-14; First posted 2019-08-21 (Actual); Results first posted 2023-10-12 (Actual); Last update posted 2023-10-12 (Actual); Status verified 2023-10

CONDITIONS: Kidney Diseases
MeSH Terms: conditions — Kidney Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Fist Assist device (all subjects) (Experimental): All study subjects will have Stage 4 or 5 Chronic Kidney Disease (CKD) that requires them to start hemodialysis. In preparation for hemodialysis, they will have an arteriovenous fistula (AVF) procedure which provides access to the veins for dialysis.
  This study is testing a device called the Fist Assist to dilate the vein in preparation for dialysis. The device is similar to a blood pressure cuff (worn around the arm and applies pressure). All study participants will wear the Fist Assist twice a day up to three months before their AVF procedure.
  Interventions: Device: Fist Assist

INTERVENTIONS:
Device: Fist Assist — The Fist Assist device works by applying pressure to the subject's arm in the area where their arteriovenous fistula will eventually be created. The device is mobile and battery powered.
  The Fist Assist device will be assigned to each enrolled subject by randomization code. All subjects will be asked to use their assigned device twice daily, for two 2-hour sessions, once in the morning and once in the evening. Patients will apply the device to the non-dominant arm above the level of the elbow, and to keep a written log to record use, complications and any problems. They will be asked to do this for 3 months, and will come in to be evaluated via study visits at Months 3, 6, 9 and 12.

SUMMARY:
This is a single center pilot study that is seeking to determine whether the use of the Fist Assist® device for 360 hours over 90 days by patients with advanced CKD prior to AVF surgery results in significant increases in cephalic vein diameters prior to AVF surgery.

DETAILED DESCRIPTION:
METHODOLOGY:

Intervention: The Fist Assist® device will be assigned to each enrolled subject by randomization code. All subjects will be asked to use their assigned device twice daily, for two 2-hour sessions, once in the morning and once in the evening. Patients will apply the device to the non-dominant arm above the level of the elbow, and to keep a written log to record use, complications and any problems.

Blood Draws: 10 mL of blood will be obtained from patients being enrolled at the time of their next routine standard of care phlebotomy. These samples will be frozen for future assays of endothelial biomarkers of nitric oxide production and venous dilation, such as asymmetric dimethyl arginine (ADMA) and its metabolites.

Doppler: Patients will undergo examination of their cephalic veins in the Nephrology Clinic, using a portable vascular ultrasound device operated by a co-investigator trained by the University of Chicago Medical Center Vascular Lab in this technique. The cephalic vein, a superficial vein originating in the wrist, is the most common vein used for AVF creation. In order to standardize these measurements, the diameter of the cephalic vein and vein wall thickness will be measured in both arms at: (a) 5 cm proximal to the styloid process of the radius, and (b) at the antecubital fossa. The diameter and thickness of the vein will be measured using a B-mode image acquired using a standard ultrasound machine with vascular probe going from outer walls per protocol. Patients will be seated with arms supported at the level of the heart on an exam table with in a room with a temperature of at least 20 degrees Celsius. A layer of at least 1 cm of gel will be applied locally to optimize the ultrasound image quality. Vascular Doppler measurements will be obtained on both arms at the time of consent (baseline), and at the conclusion of therapy. Measurements will be recorded.

Follow Up: Those who are subsequently able to undergo successful AVF creation will be followed clinically for up to 12 months.

Protocol: Informed consent will be obtained by the co-investigators using a written consent form approved by the Institutional Review Board. After informed consent is obtained, patients will receive: physical examination of both forearms; and a vascular Doppler to determine cephalic vein diameters of the nondominant arm. A 10 mL blood sample will be drawn at the next routine phlebotomy.

Patients will be asked to apply the Fist Assist® to the upper half of the non-dominant arm. Patients will be asked to use the device twice daily for two 2-hour periods, and report any complications or problems, using a log (see log attached at end of References). Patients will have follow up examinations with measurement of cephalic vein diameter at three months after enrollment.

DURATION OF STUDY: All subjects will be enrolled and treated for three months. The duration of the study including data analysis and statistical analysis is expected to be 12 months.

STATISTICAL ANALYSES: The primary outcome of interest will be the difference in the diameter of the cephalic vein between baseline (Pre) and 3 months (Post) in patients treated with the Fist Assist® device. Based on prior work, mean vein diameters at baseline are anticipated to be approximately 1.8 mm with a standard deviation of 0.5 mm,44 and investigators anticipate that the standard deviation of the change in diameter is likely to be approximately 0.75 mm.

Effect =[(DSPost)-(DSPre)]

Investigators would consider calculated effect sizes of 0.25-1.0 mm to be clinically meaningful changes that would increase the numbers of patients with vein diameters that meet commonly accepted thresholds for surgical suitability (normally 2.5-3.0 mm). Sample size calculations for a variety of effects are presented in table 1 (below), based on paired t-tests with alpha error of 0.05, standard deviation of the effect size of 0.75 mm, for power of 80% and 90%.

ELIGIBILITY:
Inclusion Criteria:

* 18 and older
* Followed in the University of Chicago Medical Center's Nephrology Clinic
* Expected to initiate hemodialysis
* Estimated Glomerular Filtration Rate (eGFR) <30 mL/min.1.73m

Exclusion criteria:

* Refusal/inability to give informed consent
* Inability to comply with trial requirements,
* Arm infections and/or skin disorders that require frequent medical attention.
* Patients with obvious scarring from IV drug use
* Previous phlebitis.
* Previous occluded arteriovenous grafts or fistulae
* Arterial aneurysms
* Arm deep vein thrombosis
* Any previous vascular surgery on the non-dominant arm.
* Limited cognitive ability
* Motor or sensory deficits in the upper arm
* Upon preliminary evaluation of the cephalic vein (measured 5 cm proximal to the styloid process of the radius, and at the antecubital fossa) there are no detectable superficial veins of at least 1.0 mm diameter, or superficial vein of more than 3.0 mm is present in this lower arm location.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2019-05-13 (Actual); Primary Completion 2022-07-27 (Actual); Study Completion 2022-07-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary Hammes, MD, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago Medical Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Fist Assist Device (All Subjects): All study subjects will have Stage 4 or 5 Chronic Kidney Disease (CKD) that requires them to start hemodialysis. In preparation for hemodialysis, they will have an arteriovenous fistula (AVF) procedure which provides access to the veins for dialysis.
  This study is testing a device called the Fist Assist to dilate the vein in preparation for dialysis. The device is similar to a blood pressure cuff (worn around the arm and applies pressure). All study participants will wear the Fist Assist twice a day up to three months before their AVF procedure.
  Fist Assist: The Fist Assist device works by applying pressure to the subject's arm in the area where their arteriovenous fistula will eventually be created. The device is mobile and battery powered.
  The Fist Assist device will be assigned to each enrolled subject by randomization code. All subjects will be asked to use their assigned device twice daily, for two 2-hour sessions, once in the morning and once in the evening. Patients will apply the device to the non-dominant arm above the level of the elbow, and to keep a written log to record use, complications and any problems. They will be asked to do this for 3 months, and will come in to be evaluated via study visits at Months 3, 6, 9 and 12.
Period: Overall Study
Arm/Group | Fist Assist Device (All Subjects)
Started | 46
Completed | 37
Not Completed | 9
Not completed — Inadequate Doppler data | 4
Not completed — Lost to Follow-up | 2
Not completed — Death | 3

BASELINE CHARACTERISTICS:
Arm/Group | Fist Assist Device (All Subjects)
Number analyzed (Participants) | 37
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.10 (12.61)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 21
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African-American | 16
  Caucasian | 6
  Other | 15

OUTCOME MEASURES:

1. Primary Outcome: Vein Diameter
Description: The primary outcome will be the difference in the vein diameter measured in millimeters with use of a vascular ultrasound device before and after Fist Assist use. The standard deviation of the change in vein diameter will be approximately 0.75mm.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: millimeters
Arm/Group | Fist Assist Device (All Subjects)
Number analyzed (Participants) | 37
millimeters
  Baseline (before) | 1.692 (0.865)
  At 3month (after) | 2.100 (0.158)
Statistical Analysis 1: Comparison: Fist Assist Device (All Subjects); Compare before and after use of Fist Assist; Test type: Equivalence — The null hypothesis is the difference is zero. Thus the equivalence margin equals zero; p = 0.012, t-test, 2 sided; Paired t-test; Mean Difference (Final Values) = 0.408, Standard Deviation 1.05

2. Secondary Outcome: AVF Creation
Description: Whether or not an arteriovenous fistula was created, as defined by a procedure performed by surgery or interventional radiology connecting an artery to a vein.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Fist Assist Device (All Subjects)
Number analyzed (Participants) | 37
Participants
  no | 20
  yes | 16
  unknown | 1

3. Secondary Outcome: AVF Maturation
Description: Whether the resultant AVF matured, as defined successful cannulation with two needles for three hemodialysis treatments.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Fist Assist Device (All Subjects)
Number analyzed (Participants) | 37
Participants
  no | 24
  yes | 12
  unknown | 1

4. Secondary Outcome: Subsequent Exposure to Central Venous Catheters
Description: The subject's subsequent exposure of patients to central venous catheters during their first year for hemodialysis. We measured the total number of patients who had exposed to central venous catheters over the first year.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Fist Assist Device (All Subjects)
Number analyzed (Participants) | 37
Participants
  no | 15
  yes | 19
  unknown | 3

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Fist Assist Device (All Subjects)
All-Cause Mortality (participants affected / at risk) | 3/46
Serious Adverse Events (participants affected / at risk) | 0/46
Other Adverse Events (participants affected / at risk) | 0/46

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-05-13): https://cdn.clinicaltrials.gov/large-docs/87/NCT04063787/Prot_SAP_000.pdf